CLINICAL TRIAL: NCT00187772
Title: Preschooler Witnesses of Domestic Violence: A Preventive Intervention Program
Brief Title: Child-Parent Psychotherapy for Preschooler Witnesses of Domestic Violence Program
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21MH059661 (NIH); R21MH059661 (NIH); IRB #HR 793-12912-06
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Domestic Violence Exposure
Keywords: domestic violence; preschoolers; trauma; intervention
MeSH Terms: conditions — Wounds and Injuries

INTERVENTIONS:
Behavioral: Child-Parent Psychotherapy (CPP)

SUMMARY:
This study will examine the efficacy of Child-Parent Psychotherapy (CPP) for the treatment of preschoolers exposed to marital violence.

DETAILED DESCRIPTION:
This study examines the efficacy of Child-Parent Psychotherapy (CPP) for the treatment of preschoolers exposed to marital violence. Multi-ethnic preschool-mother dyads from diverse socioeconomic backgrounds were randomly assigned to CPP or to a case management plus community referral for individual treatment comparison group. It was hypothesized the children who received CPP treatment would show significantly greater improvement in general symptomatology and in traumatic stress symptoms than those in the comparison group.

There is growing recognition that, contrary to the long-standing assumption that young children are impervious to environmental stresses, preschoolers exposed to violence show increased rates of disturbances in self-regulation and in emotional, social and cognitive functioning (Osofsky, 2004; Pynoos et al., 1999; van der Kolk, 2003). The present study examines the efficacy of a relationship-based treatment approach involving the child and the mother. Dyads were randomly assigned to either the Child-Parent Psychotherapy (CPP) treatment group or to a comparison group that consisted of monthly case management by an experienced Ph.D.-level clinician plus referrals for individual treatment in the community for mothers and child. We hypothesized that Child-Parent Psychotherapy would be more effective in alleviating children's traumatic stress symptoms and behavior problems because it focuses on improving the quality of the child-mother relationship and engages the mother as the child's ally in coping with the trauma. Treatment was offered for 50 weeks.

ELIGIBILITY:
Inclusion Criteria:

* child 3-5 years old
* child exposed to marital violence as confirmed by mother's report on the Conflict Tactics Scale 2 (Straus et al., 1996)
* perpetrator was not living in the home.

Exclusion Criteria:

* mother's documented abuse of the target child
* current maternal substance abuse
* homelessness
* maternal mental retardation
* maternal psychosis
* child mental retardation or autistic-spectrum disorder

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60
Dates: Start 1996-12; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Child symptomatology (CBCL)
Traumatic stress symptomatology (DC 0-3 Traumatic Stress Disorder)
Parent-Child Relationship at posttreatment and 6 month follow-up.

SECONDARY OUTCOMES:
Maternal symptomatology (Symptom Checklist Revised and Clinician Administered PTSD Scale)
Child cognitive functioning (WPPSI-R)

CONTACTS AND LOCATIONS:
Overall Officials: Alicia F. Lieberman, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- Child Trauma Research Project, San Francisco, California, United States

REFERENCES:
- [Result] Lieberman AF, Van Horn P, Ippen CG. Toward evidence-based treatment: child-parent psychotherapy with preschoolers exposed to marital violence. J Am Acad Child Adolesc Psychiatry. 2005 Dec;44(12):1241-8. doi: 10.1097/01.chi.0000181047.59702.58. PMID 16292115